CLINICAL TRIAL: NCT05724368
Title: Efficacy of Calprotectin as A Marker For the Pathogenicity of Blastocystis Infection
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Shimaa Refaey Mohamed Abd-Elal, Assistant lecturer of medical parasitology at the Faculty of Medicine, Sohag University
Other Study IDs: Soh-Med-23-01-24
Record Dates: First submitted 2023-02-02; First posted 2023-02-13 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Blastocystis Infections
Keywords: Blastocystis; Calprotectin
MeSH Terms: conditions — Blastocystis Infections

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — fecal specimens
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1: Patients with gastrointestinal symptoms and positive only for Blastocystis.
  Interventions: Diagnostic Test: Fecal Calprotectin ELISA kit
- Group 2: Patients with gastrointestinal symptoms and Blastocystis free.
  Interventions: Diagnostic Test: Fecal Calprotectin ELISA kit
- Group 3: Healthy volunteers with neither gastrointestinal symptoms nor parasitological infections.
  Interventions: Diagnostic Test: Fecal Calprotectin ELISA kit

INTERVENTIONS:
Diagnostic Test: Fecal Calprotectin ELISA kit — * Routine stool examination will be done in addition to certain concentration, staining and culture techniques.
  * Fecal calprotectin will be evaluated using ELISA kits according to the manufacturer's instructions.

SUMMARY:
Blastocystis which is commonly found in the gastro-intestinal tract, has been recognized as a non-pathogenic organism for a few decades. It has a variable distribution. A high prevalence has been reported in developing countries (22.1-100%).

In developed countries, the prevalence ranges from 0.5% to 23.1%. The high prevalence noted in developing countries is related to poor hygiene and lack of safe water and food .

DETAILED DESCRIPTION:
Blastocystis which is commonly found in the gastro-intestinal tract, has been recognized as a non-pathogenic organism for a few decades. It has a variable distribution. A high prevalence has been reported in developing countries (22.1-100%).

In developed countries, the prevalence ranges from 0.5% to 23.1%. The high prevalence noted in developing countries is related to poor hygiene and lack of safe water and food. The pathogenicity of Blastocystis is controversial because most patients carrying this parasite are asymptomatic. Several studies have considered Blastocystis sp. as a commensal micro-organism, while other results have showed the pathogenicity of the parasite.

Calprotectin (CP), a calcium-binding protein, comprises 60% of cytosolic protein found in neutrophils. Fecal calprotectin (F-CP) concentration is an indicator of neutrophil migration into the intestinal lumen and is associated with intestinal inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Patients from outpatient clinics, Sohag hospitals.

Exclusion Criteria:

* Patients taking antibiotics within the previous four weeks, and anti-parasitic drugs within the previous two weeks.

Ages: 6 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: samples will be collected from outpatients with any age & sex groups from different locations (cities and villages).
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-03 (Estimated); Primary Completion 2024-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
level of fecal calprotectin | 1 month
  Evaluation of fecal calprotectin inflammation levels of Blastocystis hominis in patients with gastrointestinal troubles as compared to patients with gastrointestinal troubles but without Blastocystis hominis

IPD SHARING:
Plan to Share IPD: Undecided